CLINICAL TRIAL: NCT06556654
Title: Evaluation of the Safety and Effectiveness of the GORE® Tissue Reinforcement for Breast Reconstruction Device (TRBR Device) When Used in the Reinforcement of Breast Reconstruction
Brief Title: Tissue Reinforcement for Breast Reconstruction (TRBR) Pivotal Clinical Study (REDEFINE)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: W.L.Gore & Associates (Industry)
Collaborators: Avania (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TBR 22-07
Record Dates: First submitted 2024-07-16; First posted 2024-08-16 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Breast Reconstruction Surgery
Keywords: breast reconstruction; post-mastectomy; tissue expander; implant based breast reconstruction; two-stage; immediate; subpectoral; prepectoral

STUDY DESIGN:
Intervention Model Description: This study is a investigational, multi-center, single-arm pivotal study to review safety outcomes of prospectively treated subjects who underwent two-stage implant-based breast reconstruction with the TRBR Device (TRBR Device group) to control subjects who underwent two-stage implant-based breast reconstruction with no mesh/ADM (Control group). Effectiveness of TRBR will be evaluated by comparing change from baseline (pre-index procedure) at 1-year post-index procedure in BREAST-Q.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Prospective Arm (Experimental): Prospectively treated subjects who undergo two-stage implant-based breast reconstruction with the TRBR Device (TRBR Device group)
  Interventions: Device: TRBR Device

INTERVENTIONS:
Device: TRBR Device — The GORE® Tissue Reinforcement for Breast Reconstruction device is intended to reinforce the soft tissue surrounding the tissue expander in preparation for the breast implant in post-mastectomy breast reconstruction

SUMMARY:
The GORE Tissue Reinforcement for Breast Reconstruction (TRBR) research study will look at breast reconstruction during mastectomy procedures. There will be two arms in this study, a Treatment Arm, where data will be collected for a new medical device called the Tissue Reinforcement for Breast Reconstruction (TRBR) Device and a Control Arm where data will be collected from subjects who have previously had surgery and received no additional tissue reinforcement in their breast reconstruction surgery. This research study will look at the safety of the Study Device and the success of the participants breast reconstruction. The Study Device is investigational, which means it has not yet been used nor approved by the FDA for this treatment. The data collected in this study will be compared to the data collected in the Control Arm.

ELIGIBILITY:
Inclusion Criteria:

1. Female subjects ≥ 22 years of age.
2. First-time breast reconstruction post-mastectomy for target breast(s).
3. Scheduled to undergo unilateral or bilateral mastectomy with immediate, two-stage, implant-based, subpectoral or prepectoral breast reconstruction after mastectomy.
4. Mastectomy performed to address breast cancer or for cancer prophylaxis.
5. An informed consent form is signed by Subject or Legally Authorized Representative (LAR).
6. Subject is capable of following protocol procedures and complying with follow-up visit requirements

Exclusion Criteria:

Baseline Exclusion Criteria

1. Subject has had a revision(s) in the target breast(s) following complications of breast augmentation, mastopexy (breast lift), or breast reduction.
2. Subject has undergone previous radiation therapy to the reconstruction site or chest wall.
3. Subject has had chemotherapy within 3 weeks prior to the index procedure.
4. Subject has been treated for a systemic infection or local infection at the surgical site within 30 days prior to index procedure.
5. Subject has a current or previous diagnosis of Methicillin-resistant Staphylococcus aureus (MRSA).
6. Subject has a BMI > 35.
7. Subject has a known diagnosis of diabetes with a HbA1c > 7.0mmol/L within 30 days of the Index procedure (i.e., TE placement).
8. Subject was a current or former tobacco/nicotine user, within 90 days prior to Index Surgery (i.e., TE placement).
9. Subject is currently taking medication (e.g., systemic steroid), which in the investigator's opinion, may increase the risk of local complications of breast reconstruction.
10. Subject has other medical, social, or psychological conditions which could interfere with provision of informed consent, completion of tests, therapy, or follow-up.
11. Subject is currently participating in or planning to participate in another investigational drug, biologic or medical device study that may interfere with compliance of TBR 22-07 study requirements or may confound TBR 22-07 study data/outcomes.
12. Subject requires a surgical technique requiring flap (autologous tissue).
13. Subject is pregnant or lactating at the time of the index procedure (i.e., TE placement) or is planning to become pregnant prior to the Exchange procedure. Intraoperative Index Procedure Exclusion
14. Based on investigator's opinion, subject has unsuitable tissue integrity for immediate 2-stage breast reconstruction or is no longer a candidate to receive the TRBR Device (will be recorded as a screen failure).
15. Subject receives an Acellular Dermal Matrix (ADM) or mesh that is not the TRBR Device in the target breast(s)

Min Age: 22 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female at birth
Enrollment: 180 (Estimated)
Dates: Start 2025-04-09 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Absence of device- or procedure-related major adverse events (MAEs) | 1 year post index procedure
  Require rehospitalization or reoperation

SECONDARY OUTCOMES:
BREAST-Q Physical Well Being | 1-year post-index procedure.
  Chest Score change from baseline (pre-index procedure).

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Hammond, MD, Principal Investigator — Partners in Plastic Surgery of West Michigan
Locations (20):
- United States (20):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - University of Arizona, Tucson, Arizona
  - The Regents of the University of California, Irvine, California
  - Cedars-Sinai Plastic and Reconstruction Surgery, Los Angeles, California
  - Riverside University Health System-Medical Center, Moreno Valley, California
  - Mayo Clinic Florida, Jacksonville, Florida
  - Endeavor Health (Northshore University HealthSystem Research Institute), Evanston, Illinois
  - Northwestern University, Evanston, Illinois
  - BR Hope LLC, Wichita, Kansas
  - The Johns Hopkins University, Baltimore, Maryland
  - Corewell Health Research Institute, Grand Rapids, Michigan
  - University of Mississippi, Jackson, Mississippi
  - The Board of Regents of the University of Nebraska, Omaha, Nebraska
  - The Joan and Sanford I. Weill Medical College of Cornell University, New York, New York
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - The Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - The University of Washington Medical Center, Seattle, Washington
  - The Board of Regents of the University of Wisconsin System, Madison, Wisconsin
  - The Medical College of Wisconsin, Inc., Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No